CLINICAL TRIAL: NCT01428687
Title: Increasing Sleep Duration: A Novel Approach to Weight Control
Brief Title: Short Term Effects of Increasing Sleep Duration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Principal Investigator, Rena R. Wing, Professor of Psychiatry and Human Behavior, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U01CA150387 - Study 2; U01CA150387 (NIH)
Record Dates: First submitted 2011-09-01; First posted 2011-09-05 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Overweight and Obesity
Keywords: Weight loss; Sleep duration
MeSH Terms: conditions — Overweight; Obesity; Weight Loss | interventions — Sleep Duration; Sleep

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Increase Sleep Gradually (Active Comparator): Subjects in this condition are taught to increase their sleep by 30 minutes per night during week 1 of the intervention; 60 minutes during week 2; and 90 minutes during week 3. Following the sleep intervention, these participants receive a standard behavioral with loss intervention.
  Interventions: Behavioral: Sleep Duration
- Increase Sleep Immediately (Active Comparator): Subjects in this condition are taught to increase their sleep by 90 minutes per night starting in week 1. Following the sleep intervention, these participants receive a standard behavioral with loss intervention.
  Interventions: Behavioral: Sleep Duration
- No Intervention: Control Group (Active Comparator): This group is told to make no changes in their sleep habits. Following the sleep intervention, these participants receive a standard behavioral with loss intervention.
  Interventions: Behavioral: No change in sleep

INTERVENTIONS:
Behavioral: Sleep Duration — Subjects are taught sleep hygiene strategies to increase their sleep; they record their sleep in a diary and wear an actigraph and call in their sleep to the office each day.
  Arms: Increase Sleep Gradually; Increase Sleep Immediately
Behavioral: No change in sleep — This group is taught to maintain their current sleep habits.
  Arms: No Intervention: Control Group

SUMMARY:
A series of studies are proposed to develop an intervention to increase sleep duration and study the effects on eating, exercise, and weight control. The hypothesis is that increasing sleep duration will help improve weight loss and maintenance.

DETAILED DESCRIPTION:
Study 1 is conducted in a sleep laboratory. Participants sleep short duration (approximately four hours per night) on one weekend and long duration (approximately nine hours per night) on another weekend.

Study 2 is examining ways to increase sleep duration in overweight individuals with short sleep and examining the effects on short term weight loss.

Study 3 is comparing a standard weight loss program with a novel Sleep+Weight Loss intervention.

ELIGIBILITY:
Inclusion Criteria:

* age 25 to 45;
* BMI 25 to 50;
* healthy;
* sleep 6.5 hours or less per night

Exclusion Criteria:

* use of sleep medications;
* sleep apnea;
* third shift worker

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Sleep Duration | 4 weeks
  Participants with verified short sleep are taught to increase their sleep either gradually or immediately. These two groups are compared to a control group who makes no changes in their sleep. The primary outcome is sleep duration per night as determined by actigraphy.

SECONDARY OUTCOMES:
Eating Behavior | 4 weeks
  24-hour recalls are used to estimate dietary intake at baseline and after 4 weeks of sleep intervention.
Physical Activity | 4 weeks
  Objective measures of physical activity are obtained before and after the 4-week sleep intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Rena R. Wing, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- Weight Control & Diabetes Research Center, Providence, Rhode Island, United States